CLINICAL TRIAL: NCT00004925
Title: Phase I/II Study of TLC D-99 Plus Herceptin as First or Second Line Therapy for Patients With Locally Advanced Inflammatory or Metastatic Breast Cancer
Brief Title: Liposomal Doxorubicin and Trastuzumab in Treating Women With Locally Advanced, Inflammatory, or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-054; CDR0000067609 (Registry Identifier: PDQ (Physician Data Query)); LIPO-D9905; NCI-G00-1684
Record Dates: First submitted 2000-03-07; First posted 2003-05-14 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; stage IIIB breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Trastuzumab

INTERVENTIONS:
Biological: trastuzumab
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I/II trial to study the effectiveness of liposomal doxorubicin and trastuzumab in treating women who have locally advanced, inflammatory, or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety, especially the cardiac safety, of doxorubicin HCl liposome and trastuzumab (Herceptin) as first- or second-line therapy in women with metastatic, inflammatory, or locally advanced breast cancer.

OUTLINE: Patients are stratified according to prior anthracycline therapy (yes vs no).

Patients receive doxorubicin HCl liposome IV over 1 hour followed 30 minutes later by trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, and 15. Treatment continues every 21 days in the absence of unacceptable toxicity or disease progression.

Patients are followed for at least 3 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced, inflammatory, or metastatic adenocarcinoma of the breast that has been treated with no more than 1 prior systemic cytotoxic regimen
* Overexpression of HER2 protein (2+ or 3+)
* Evaluable disease
* History of brain metastases allowed if off steroids and asymptomatic, with a 3 month or greater interval since last dose of brain irradiation, and no evidence of progression
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)

Renal:

* AST or ALT no greater than 4 times ULN

Cardiovascular:

* Adequate cardiac function
* LVEF at least 50% predicted or lower limit of normal

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent medical or psychological condition that would preclude study compliance
* No history of hypersensitivity to anthracyclines, eggs, or egg products

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior trastuzumab (Herceptin) allowed

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior antineoplastic therapy
* No more than 1 prior systemic cytotoxic regimen for locally advanced, metastatic, or inflammatory breast cancer
* No prior anthracyclines greater than 240 mg/m2
* No other concurrent antineoplastic agents
* No concurrent treatment with other liposomal products other than doxorubicin HCl liposome

Endocrine therapy:

* See Disease Characteristics
* At least 3 weeks since prior hormonal agents
* No concurrent hormonal therapy

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Other:

* At least 3 weeks since other prior investigational drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Theodoulou, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Theodoulou M, Batist G, Campos S, Winer E, Welles L, Hudis C. Phase I study of nonpegylated liposomal doxorubicin plus trastuzumab in patients with HER2-positive breast cancer. Clin Breast Cancer. 2009 May;9(2):101-7. doi: 10.3816/CBC.2009.n.019. PMID 19433391